CLINICAL TRIAL: NCT03875729
Title: Phase 3 Randomized Double-Blind Multinational Placebo-Controlled Study to Evaluate Efficacy and Safety of Teplizumab, a Humanized Fc Receptor (FcR) Non-Binding Anti-cluster of Differentiation 3 (CD3) Monoclonal Antibody, in Children and Adolescents With Newly Diagnosed Type 1 Diabetes
Brief Title: Recent-Onset Type 1 Diabetes Trial Evaluating Efficacy and Safety of Teplizumab
Acronym: PROTECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Provention Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRV-031-001
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1D, type 1 diabetes, recent-onset T1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Intervention Model Description: Phase 3, randomized, double-blind, placebo-controlled, multinational, multicenter study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Teplizumab (Experimental): Teplizumab was administered via intravenous infusion in two courses, with the first course starting on Day 1 (Week 1) and the second course approximately 6 months later at Day 182 (Week 26). Participants who were unable to receive the second 12-day course due to COronaVIrus Disease of 2019 (COVID-19) pandemic restrictions were given the second course at approximately 12 months (Week 52 visit). Each course of treatment included daily infusions for 12 days.
  Each course included:
  * Day 1: 106 μg/m^2
  * Day 2: 425 μg/m^2
  * Days 3-12: 850 μg/m^2 Total per course: 9.0 mg/m^2 The doses of study drug were calculated based on the participant's body surface area (BSA) measured on the first day of each treatment course.
  Interventions: Biological: teplizumab
- Placebo (Placebo Comparator): Placebo was administered via intravenous infusion in two courses, with the first course starting on Day 1 (Week 1) and the second course approximately 6 months later at Day 182 (Week 26). Participants who were unable to receive the second 12-day course due to COronaVIrus Disease of 2019 (COVID-19) pandemic restrictions were given the second course at approximately 12 months (Week 52 visit). Each course of treatment included daily infusions for 12 days.
  The placebo solution consisted of the same formulation as the study drug but without teplizumab. Placebo was administered in the same dose volume and by the same treatment schedule as the active drug.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: teplizumab — Treatment
  Arms: Teplizumab
Biological: Placebo — Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether teplizumab slows the loss of β cells and preserves β cell function in children and adolescent 8-17 years old who have been diagnosed with T1D in the previous 6 weeks..

Subjects will receive two courses of either teplizumab or placebo treatment 6 months apart.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, multinational, multi-center study to evaluate the efficacy and safety of teplizumab, a humanized, anti-CD3 monoclonal antibody, in children and adolescents ages 8 through 17 recently diagnosed with type 1 diabetes (within 6 weeks of diagnosis). Approximately 300 participants will be randomized at a ratio of 2:1 to either the teplizumab group or the placebo group.

Teplizumab or matching placebo will be administered in two courses 6 months apart. Each course of treatment will include daily infusions for 12 days. The total study duration for each participant will be up to 86 weeks.

The primary objective is to determine whether two courses of teplizumab administered 6 months apart slows the loss of β cells and preserves β cell function over 18 months (78 weeks) in children and adolescents 8-17 years old who have been diagnosed with T1D in the previous 6 weeks.

The secondary objectives are to evaluate improvements in key clinical parameters of diabetes management, to determine the safety and tolerability of teplizumab, and to evaluate the pharmacokinetics (PK) and immunogenicity of teplizumab

ELIGIBILITY:
Inclusion Criteria:

1. Is 8 to 17 years of age, inclusive, at the time of randomization/initiation of study drug administration.
2. Has received a diagnosis of type 1 diabetes (T1D) according to the criteria from the American Diabetes Association.
3. Is able to be randomized and initiate study drug within 6 weeks (42 days) of the formal T1D diagnosis.
4. Has a peak stimulated C-peptide of ≥0.2 pmol/mL from a mixed meal tolerance test (MMTT) at screening.
5. Has a positive result on testing for T1D-related autoantibodies.

Exclusion Criteria:

1. Has any autoimmune disease other than T1D with the exception of stable thyroid or celiac disease.
2. Has an active infection and/or fever.
3. Has a history of or serologic evidence at screening of current or past infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
4. An individual who has a medical, psychological or social condition that, in the opinion of the Principal Investigator, would interfere with safe and proper completion of the trial.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 328 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Provention Bio, Inc.
Locations (62):
- United States (34):
  - Rady Children's Hospital-San Diego (Site 004), San Diego, California
  - UCSF Medical Center (Site 001), San Francisco, California
  - Diablo Clinical Research, Inc. (Site 002), Walnut Creek, California
  - University of Colorado-Barbara Davis Center for Childhood Diabetes (Site 005), Aurora, Colorado
  - Yale University of Medicine (Site 020), New Haven, Connecticut
  - UF Clinical and Translation Research Building (Site 015), Gainesville, Florida
  - Nemours Children's Specialty Care-Endocrinology (Site 047), Jacksonville, Florida
  - University of Miami Health System (Site 028), Miami, Florida
  - All Children's Hospital-Johns Hopkins Medicine (Site 048), St. Petersburg, Florida
  - University of South Florida Diabetes and Endocrinology Center (Site 011), Tampa, Florida
  - Atlanta Diabetes Associates (Site 009), Atlanta, Georgia
  - Centricity Research (Site 006), Columbus, Georgia
  - St. Luke's Children's Endocrinology (Site 052), Boise, Idaho
  - Rocky Mountain Diabetes and Osteoporosis Center (Site 007), Idaho Falls, Idaho
  - University of Chicago Medical Center (Site 017), Chicago, Illinois
  - Indiana University Hospital and Riley Hospital for Children (Site 014), Indianapolis, Indiana
  - U. Iowa Children's Hospital (Site 023), Iowa City, Iowa
  - Capital Diabetes & Endocrine Associates (Site 029), Camp Springs, Maryland
  - Baystate Pediatric Endocrinology & Diabetes (Site 040), Springfield, Massachusetts
  - U. Minnesota Health Clinical Research Unit (Site 031), Minneapolis, Minnesota
  - Children's Mercy Hospitals & Clinics (Site 026), Kansas City, Missouri
  - Washington University School of Medicine (Site 018), St Louis, Missouri
  - Women and Children's Hospital of Buffalo (Site 010), Buffalo, New York
  - UNC Hospitals Children's Specialty Clinic (Site 038), Chapel Hill, North Carolina
  - Rainbow Babies & Children's Hospital (Site 049), Cleveland, Ohio
  - Cleveland Clinic (Site 051), Cleveland, Ohio
  - Endocrinology Service Northwest, LLC (Site 034), Bend, Oregon
  - Childrens Hospital of Philadelphia - Endocrinology (Site 021), Philadelphia, Pennsylvania
  - Sanford Diabetes and Thyroiid Clinical (Site 013), Sioux Falls, South Dakota
  - AM Diabetes & Endocrinology Center (Site 008), Bartlett, Tennessee
  - Vanderbilt University Medical Center (Site 024), Nashville, Tennessee
  - Children's Medical Center Dallas (Site 033), Dallas, Texas
  - Benaroya Research Institute at Virginia Mason (Site 016), Seattle, Washington
  - MultiCare Institute for Research & Innovation (Site 003), Tacoma, Washington
- Belgium (3):
  - UZ Brussel - Campus Jette (Site 202), Brussels, Brussels Capital
  - UZ Gent (Site 206), Ghent, Oost-Vlaanderen
  - CHU UCL Namur, site Clinique Sainte-Elisabeth (Site 205), Namur
- Canada (3):
  - Alberta Diabetes Institute Clinical Research Unit Li Ka Shing Centre for Health Research Innovation (Site 103), Edmonton, Alberta
  - BC Diabetes (Site 102), Vancouver, British Columbia
  - Montreal Children's Hospital-McGill (Site 101), Montreal, Quebec
- Fakultni nemocnice v Motole (Site 301), Prague, Czechia
- France (7):
  - Hopitaux Pediatriques de Nice CHU-Lenval service de diabetologie et d'endocrinologia (Site 508), Nice, Alpes-Maritimes
  - CHU Hopital de la Timone-Hopital d'Enfants (Site 512), Marseille, Bouces-du-Rhone
  - CHU DIJON hopital d'enfant (Site 504), Dijon, cote-d'Or
  - Centre Hospitalier Regional (CHR) d'Orleans-Service de pediatrie (Site 513), Orléans, Loiret
  - Groupe hospitalier Est-Hopital Femme, Mere, Enfant (Site 509), Bron, Rhone
  - Centre hospitalier de Pau (Site 501), Pau
  - Groupe Hospitalier Necker Enfants Malades (site 502), Paris, Île-de-France Region
- Germany (6):
  - Universitätsklinikum Freiburg (Site 603), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg (Site 608), Heidelberg, Baden-Wurtternberg
  - Universitätsklinikum Augsburg (Site 606), Augsburg, Bayem
  - Evangelisches Klinikum Bethel Kinderklinik (Site 602), Bielefeld, North Rhine-Westphalia
  - Universitatsklinikum Carl Gustav Carus (Site 601), Dresden, Sachson
  - Kinderkrankenhaus Auf Der Bult (Site 604), Hanover
- Békés Megyei Központi Kórház Pándy Kálmán Tagkórház ( Site 705), Gyula, Hungary
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu (Site 804), Warsaw, Masovian Voivodeship
  - Instytut Diabetologii Sp. z o.o. (Site 802), Warsaw
  - Instytut "Pomnik - Centrum Zdrowia Dziecka" (Site 801), Warsaw
  - Uniwersyteckie Centrum Kliniczne (Site 803), Warsaw
- United Kingdom (3):
  - Northwick Park Hospital - Paediatrics (site 904), London, City of London
  - Cardiff and Vale NHS Trust - University Hospital of Wales (Site 902), Cardiff
  - Sheffield Children's NHS Foundation Trust Western Bank (Site 903), Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient levels data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After drug approval
Access Criteria: Qualified researchers
URL: http://Vivli.org

REFERENCES:
- [Result] Ramos EL, Dayan CM, Chatenoud L, Sumnik Z, Simmons KM, Szypowska A, Gitelman SE, Knecht LA, Niemoeller E, Tian W, Herold KC; PROTECT Study Investigators. Teplizumab and beta-Cell Function in Newly Diagnosed Type 1 Diabetes. N Engl J Med. 2023 Dec 7;389(23):2151-2161. doi: 10.1056/NEJMoa2308743. Epub 2023 Oct 18. PMID 37861217
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417
- [Derived] Novograd J, Frishman WH. Teplizumab Therapy to Delay the Onset of Type 1 Diabetes. Cardiol Rev. 2024 Nov-Dec 01;32(6):572-576. doi: 10.1097/CRD.0000000000000563. Epub 2023 May 9. PMID 37158990
- See also: New England Journal of Medicine publication of the study results — http://pubmed.ncbi.nlm.nih.gov/37861217/
- Available data/document: Individual Participant Data Set — https://www.vivli.org/ — Qualified researchers can submit a research proposal that includes specific information about the purpose of the research, the objectives, the analysis plan, the publication plan, etc. Qualified researchers may request access to patient level data and related study documents. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on April 5, 2019, and the last participant was enrolled on November 4, 2021.
Pre-assignment Details: Of 422 assessed for eligibility, 328 met inclusion criteria and were randomized to treatment.
Groups:
- Placebo: Placebo: Control
  Placebo was administered via intravenous infusion in two courses, with the first course starting on Day 1 (Week 1) and the second course approximately 6 months later at Day 182 (Week 26). Participants who were unable to receive the second 12-day course due to COronaVIrus Disease of 2019 (COVID-19) pandemic restrictions were given the second course at approximately 12 months (Week 52) in a modified dosing schedule. Each course of treatment included daily infusions for 12 days.
  The placebo solution consisted of the same formulation as the study drug but without teplizumab.
  Placebo was administered in the same dose volume and by the same treatment schedule as the active drug.
- Teplizumab: Teplizumab: Treatment
  Teplizumab was administered via intravenous infusion in two courses, with the first course starting on Day 1 (Week 1) and the second course approximately 6 months later at Day 182 (Week 26). Participants who were unable to receive the second 12-day course due to COronaVIrus Disease of 2019 (COVID-19) pandemic restrictions were given the second course at approximately 12 months (Week 52) in a modified dosing schedule. Each course of treatment included daily infusions for 12 days.
  Each course included:
  * Day 1: 106 μg/m^2
  * Day 2: 425 μg/m^2
  * Days 3-12: 850 μg/m^2 Total per course: 9.0 mg/m^2 The doses of study drug were calculated based on the participant's body surface area (BSA) measured on the first day of each treatment course.
Period: Overall Study
Arm/Group | Placebo | Teplizumab
Started | 111 | 217
Completed | 101 | 195
Not Completed | 10 | 22
Not completed — Adverse Event | 0 | 5
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 0 | 5
Not completed — Personal reasons | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Teplizumab | Total
Number analyzed (Participants) | 111 | 217 | 328
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 111 | 217 | 328
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (2.55) | 12.0 (2.53) | 12.1 (2.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 98 | 140
  Male | 69 | 119 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 14 | 18
  Not Hispanic or Latino | 101 | 193 | 294
  Unknown or Not Reported | 6 | 10 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 94 | 189 | 283
  Black or African American | 6 | 5 | 11
  Asian | 3 | 4 | 7
  American Indian or Alaskan Native | 0 | 1 | 1
  Native Hawiian or Other Pacific Islander | 1 | 0 | 1
  Multiple | 0 | 6 | 6
  Other | 1 | 4 | 5
  Not reported | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 13 | 20
  Belgium | 4 | 1 | 5
  United States | 56 | 126 | 182
  Czechia | 10 | 17 | 27
  Poland | 15 | 33 | 48
  United Kingdom | 6 | 6 | 12
  France | 5 | 9 | 14
  Germany | 8 | 12 | 20
Peak C-peptide at screening [Count of Participants; unit: Participants]
  0.2 - 0.7 pmol/mL | 47 | 91 | 138
  >0.7 pmol/mL | 64 | 126 | 190
Age group at randomization [Count of Participants; unit: Participants]
  8 - 12 years | 62 | 120 | 182
  >12 - 17 years | 49 | 97 | 146
Number of positive type 1 diabetes (T1D) autoantibodies [Count of Participants; unit: Participants]
  None | 0 | 1 | 1
  One | 3 | 10 | 13
  Two | 13 | 38 | 51
  Three | 30 | 47 | 77
  Four | 39 | 66 | 105
  Five | 26 | 55 | 81
History of diabetic ketoacidosis (DKA) [Count of Participants; unit: Participants]
  Yes | 4 | 0 | 4
  No | 107 | 217 | 324
Human leukocyte antigen (HLA) genotyping - DR3 [Count of Participants; unit: Participants] — Population: Populations differs due to missing values.
  Participants
    number analyzed (Participants) | 109 | 215 | 324
    Positive | 56 | 96 | 152
    Negative | 53 | 119 | 172
Human leukocyte antigen (HLA) genotyping - DR4 [Count of Participants; unit: Participants] — Population: Populations differs due to missing values.
  Participants
    number analyzed (Participants) | 109 | 215 | 324
    Positive | 75 | 137 | 212
    Negative | 34 | 78 | 112
Anti-glutamic acid decarboxylase 65 (GAD65) autoantibody [Count of Participants; unit: Participants]
  Positive | 96 | 183 | 279
  Negative | 15 | 34 | 49
Anti-islet antigen 2 (IA-2) autoantibody [Count of Participants; unit: Participants]
  Positive | 87 | 165 | 252
  Negative | 24 | 52 | 76
Anti-zinc transporter 8 (ZnT8) autoantibody [Count of Participants; unit: Participants]
  Positive | 83 | 162 | 245
  Negative | 28 | 55 | 83
Anti-insulin autoantibody [Count of Participants; unit: Participants]
  Positive | 85 | 144 | 229
  Negative | 26 | 73 | 99
Anti-islet cell cytoplasmic antibody (ICA) [Count of Participants; unit: Participants]
  Positive | 54 | 112 | 166
  Negative | 57 | 105 | 162
Height [Mean (Standard Deviation); unit: cm] | 158.48 (14.977) | 155.35 (15.358) | 156.41 (15.279)
Weight [Mean (Standard Deviation); unit: kg] | 49.19 (15.889) | 46.68 (14.992) | 47.53 (15.323)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 19.063 (3.6415) | 18.868 (3.4517) | 18.934 (3.5127)
Body mass index (BMI) z-score [Mean (Standard Deviation); unit: z-score] — The body mass index (BMI) z-score is a measure of the relative BMI adjusted for child's age and sex and describes the distance the BMI measurement falls from the mean in standard deviation units. A z-score of 0 represents the mean BMI for that age and sex, and a positive score indicates a BMI is higher than the mean, and a negative z-score indicates a BMI is lower than the mean. Z-scores were derived using the growth chart from the general population (e.g., Centers for Disease Control and Prevention (CDC) Growth Charts, https://www.cdc.gov/growthcharts/clinical_charts.htm).
  z-score | 0.0557 (1.0957) | 0.0627 (1.0723) | 0.0603 (1.0786)
C-peptide area under concentration-time curve standardized by mixed meal tolerance test duration [Mean (Standard Deviation); unit: pmol/mL] — The area under concentration-time curve (AUC) of C-peptide was measured after a 4-hour (4h) mixed meal tolerance test (MMTT). The AUC was computed using the trapezoidal rule and standardized by the duration of the MMTT test, i.e., AUC was divided by the last blood sample collection time (240 minutes or the last collection time for 4h MMTT).
  pmol/mL | 0.7237 (0.3190) | 0.7445 (0.3653) | 0.7375 (0.3499)
Insulin use [Mean (Standard Deviation); unit: U/kg/day] — Insulin use at baseline was calculated as the average daily use for participants who had at least 3 days of data recorded on the insulin diary before the start of the study. Population: Insulin use at baseline was not calculated for participants who did not have at least 3 days of data recorded on the insulin diary before the start of the study.
  U/kg/day
    number analyzed (Participants) | 63 | 126 | 189
    (all) | 0.383 (0.2535) | 0.447 (0.3093) | 0.426 (0.2928)
Glycated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycated hemoglobin] — Population: Population differs due to missing value for one participant.
  Percentage of glycated hemoglobin
    number analyzed (Participants) | 110 | 217 | 327
    (all) | 9.18 (1.918) | 8.90 (1.729) | 9.00 (1.797)
Time from type 1 diabetes (T1D) diagnosis to randomization [Mean (Standard Deviation); unit: weeks] | 5.20 (0.812) | 5.37 (0.730) | 5.31 (0.762)

OUTCOME MEASURES:

1. Primary Outcome: Change in C-peptide ln(AUC+1) Standardized by Duration of the Mixed Meal Tolerance Test (MMTT)
Description: The area under the concentration-time curve (AUC) of C-peptide was measured after a 4-hour mixed meal tolerance test (MMTT) and is a measure of endogenous insulin production and β cell function. The AUC was computed using the trapezoidal rule and standardized by the duration of the MMTT test, i.e., AUC was divided by the last blood sample collection time (240 minutes or the last collection time for 4h MMTT).
Time Frame: Baseline to Week 78
Population: Intent-to-treat (ITT) and Per Protocol (PP). The main reason participants were excluded from the PP population was for treatment compliance <80% (15 of 16 excluded participants in the placebo group and 32 of 37 in the teplizumab group). Other reasons included took prohibited medication (1 in placebo group, 3 in teplizumab group), received incorrect treatment (2 in teplizumab group), and pregnancy (1 in teplizumab group).
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Placebo | Teplizumab
Number analyzed (Participants) | 111 | 217
pmol/mL
  Intent-to-treat | -0.2112 [-0.2437 to -0.1786] | -0.0859 [-0.1090 to -0.0628]
  Per Protocol: number analyzed (Participants) | 95 | 180
  Per Protocol | -0.2185 [-0.2501 to -0.1869] | -0.0800 [-0.1030 to -0.0570]
Statistical Analysis 1: Comparison: Placebo vs Teplizumab; This study was designed to show a difference of at least a 40% in C-peptide response between teplizumab and placebo. In geometric means, this translates to a value of (1.4×0.28) = 0.392. Consequently, approximately 300 participants were planned for enrollment, assuming 2-sided α=0.05, 90% power, 2:1 randomization, and a 10% dropout rate; Test type: Superiority; p < 0.001, ANCOVA — ITT: The ANCOVA model included treatment, age group at randomization, and baseline C-peptide ln(AUC+1) as independent variables. Missing data at Week 78 were multiply imputed using pattern-mixture model under the missing not at random assumption; Mean Difference (Net) = 0.1253, 95% CI 2-sided [0.0852 to 0.1653] — Least squares mean (LSmean) difference = Teplizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Teplizumab; Test type: Superiority; p < 0.001, ANCOVA — PP: The ANCOVA model included treatment, age group at randomization, and baseline C-peptide ln(AUC+1) as independent variables. Missing data at Week 78 were multiply imputed using a pattern-mixture model under the missing not at random assumption; Mean Difference (Net) = 0.1385, 95% CI 2-sided [0.0994 to 0.1776] — Least squares mean (LSmean) difference = teplizumab - placebo

2. Secondary Outcome: Average Daily Exogenous Insulin Use
Description: The average daily insulin use was calculated based on participants who have at least 3 days of insulin use recorded in the dairy for the Week 78 visit.
Time Frame: Week 78
Population: Intent-to-treat and Per Protocol
Measure: Least Squares Mean (95% Confidence Interval); unit: Units/kg/day
Arm/Group | Placebo | Teplizumab
Number analyzed (Participants) | 111 | 217
Units/kg/day
  Intent-to-treat | 0.593 [0.470 to 0.716] | 0.463 [0.363 to 0.562]
  Per Protocol: number analyzed (Participants) | 95 | 180
  Per Protocol | 0.613 [0.538 to 0.687] | 0.446 [0.390 to 0.502]
Statistical Analysis 1: Comparison: Placebo vs Teplizumab; Test type: Superiority; p = 0.085, ANCOVA — ITT: ANCOVA model included treatment, age group at randomization, and screening peak C-peptide category as independent variables. Missing data at Week 78 were multiply imputed using a pattern-mixture model under the missing not at random assumption; Mean Difference (Final Values) = -0.131, 95% CI 2-sided [-0.280 to 0.018] — LSmean difference = teplizumab - placebo
Statistical Analysis 2: Comparison: Placebo vs Teplizumab; Test type: Superiority; p < 0.001, ANCOVA — PP: ANCOVA model included treatment, age group at randomization, and screening peak C-peptide category as independent variables. Missing data at Week 78 were multiply imputed using a pattern-mixture model under the missing not at random assumption; Mean Difference (Final Values) = -0.167, 95% CI 2-sided [-0.256 to -0.078] — LSmean difference = teplizumab - placebo

3. Secondary Outcome: Change in Glycated Hemoglobin (HbA1c) Levels (%)
Description: Change in percentage (%) glycated hemoglobin (HbA1c)
Time Frame: Baseline to Week 78
Population: Intent-to-treat and Per Protocol
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of glycated hemoglobin
Arm/Group | Placebo | Teplizumab
Number analyzed (Participants) | 111 | 217
Percentage of glycated hemoglobin
  Intent-to-treat | -1.89 [-2.16 to -1.62] | -1.98 [-2.17 to -1.78]
  Per Protocol: number analyzed (Participants) | 95 | 180
  Per Protocol | -1.94 [-2.21 to -1.67] | -2.07 [-2.27 to -1.87]
Statistical Analysis 1: Comparison: Placebo vs Teplizumab; Test type: Superiority; p = 0.606, ANCOVA — ITT: ANCOVA model included treatment, age group at randomization, screening peak C-peptide category, baseline HbA1c as independent variables. Missing data were multiply imputed using a pattern-mixture model under the missing not at random assumption; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.42 to 0.24]
Statistical Analysis 2: Comparison: Placebo vs Teplizumab; Test type: Superiority; p = 0.454, ANCOVA — PP: ANOVA model included treatment, age group at randomization, screening peak C-peptide category, baseline HbA1c as independent variables. Missing data were multiply imputed using a pattern-mixture model under the missing not at random assumption; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.46 to 0.20] — LSmean difference = teplizumab - placebo

4. Secondary Outcome: Time in Range for Glycemia Control
Description: Time in range (%) for glycemia control was assessed using Continuous Glucose Monitoring (CGM). Time in range was defined as daily average percentage of time a participant's glucose is >= 70 mg/dL and <=180 mg/dL. Time in range was calculated based on participants who had at least 3 days of CGM data recorded for Week 78 visit with a range of at least 8 hours on a given day.
Time Frame: Week 78
Population: Intent-to-treat and Per Protocol
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of time in range
Arm/Group | Placebo | Teplizumab
Number analyzed (Participants) | 111 | 217
Percentage of time in range
  Intent-to-treat | 62.65 [57.38 to 67.92] | 67.36 [63.70 to 71.03]
  Per Protocol: number analyzed (Participants) | 95 | 180
  Per Protocol | 61.44 [56.50 to 66.38] | 67.61 [64.09 to 71.14]
Statistical Analysis 1: Comparison: Placebo vs Teplizumab; Test type: Superiority; p = 0.151, ANCOVA — ITT: The ANCOVA model included treatment, age group at randomization, and screening peak C-peptide category as independent variables. Missing data were multiply imputed using a pattern-mixture model under the missing not at random assumption; Mean Difference (Final Values) = 4.71, 95% CI 2-sided [-1.72 to 11.15] — LSmean difference = teplizumab - placebo
Statistical Analysis 2: Comparison: Placebo vs Teplizumab; Test type: Superiority; p = 0.045, ANCOVA — PP: The ANCOVA model included treatment, age group at randomization, and screening peak C-peptide category as independent variables. Missing data were multiply imputed using a pattern-mixture model under the missing not at random assumption; Mean Difference (Final Values) = 6.17, 95% CI 2-sided [0.13 to 12.22] — LSmean difference = teplizumab - placebo

5. Secondary Outcome: Rate of Clinically Important Hypoglycemic Events
Description: Rate = clinically important hypoglycemic events/patient-year. A clinically important episode was defined as a blood glucose value of <54 mg/dL (3.0 mmol/L) (i.e., Level 2 Hypoglycemia, International Hypoglycemia Study Group, 2017) or a hypoglycemia event of severe cognitive impairment requiring external assistance (such as seizure, syncope, severe confusion with or without a confirmatory low blood glucose reading) (i.e., Level 3 Hypoglycemia, International Hypoglycemia Study Group 2017). Event rate was calculated for each participant as number of events / total study follow-up time. Total study follow-up time was calculated as (the date of last study contact - the first dose date + 1)/365.25. The summary is based on the data reported post-baseline in the Hypoglycemic Events Electronic Diary (eDiary).
Time Frame: During the entire study (from the first dose to the last study contact, up to 78 Weeks)
Population: Intent-to-treat and Per Protocol
Measure: Mean (95% Confidence Interval); unit: Events/patient-year
Arm/Group | Placebo | Teplizumab
Number analyzed (Participants) | 111 | 217
Events/patient-year
  Intent-to-treat | 4.24 [3.06 to 5.89] | 4.68 [3.70 to 5.91]
  Per protocol: number analyzed (Participants) | 95 | 180
  Per protocol | 4.63 [3.31 to 6.49] | 5.04 [3.94 to 6.44]
Statistical Analysis 1: Comparison: Placebo vs Teplizumab; Test type: Superiority; p = 0.634, Negative binomial regression model — ITT: Estimates and p-values were obtained from a negative binomial regression model using rate of hypoglycemic episodes as dependent variable and treatment, age group at randomization, and screening peak C-peptide category as independent variables; Rate ratio = 1.10, 95% CI 2-sided [0.74 to 1.64] — Rate ratio = teplizumab / placebo
Statistical Analysis 2: Comparison: Placebo vs Teplizumab; Test type: Superiority; p = 0.690, Rate ratio — PP: Estimates and p-values were obtained from a negative binomial regression model using rate of hypoglycemic episodes as dependent variable and treatment age group at randomization, and screening peak C-peptide category as independent variables; Rate ratio = 1.09, 95% CI 2-sided [0.72 to 1.65] — Rate ratio = teplizumab / placebo

6. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: AESIs are defined in the protocol and categories in the statistical analysis plan. Participants with multiple events are counted only once for each preferred term and category.
Time Frame: During the entire study (from the first dose to the last study contact, up to 78 Weeks)
Population: Safety population = all randomized study participants receiving any exposure to study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Teplizumab
Number analyzed (Participants) | 111 | 217
Participants
  Treatment-emergent AESI | 24 | 63
  Participants with at least one >= grade 3 infection | 2 | 1
  Participants with at least one acute mononucleosis-like illness | 3 | 17
  Participants with at least one lymphoma or other malignancy, including benign tumors | 1 | 2
  Participants with at least one instance of severe hypoglycemic event | 18 | 29
  Participants with at least one >=grade 3 liver function abnormality | 0 | 8
  Participants with at least one >= grade 3 thrombocytopenia | 0 | 0
  Participants with at least one >= grade 3 neutropenia | 0 | 7
  Participants with at least one >= grade 4 allergic/hypersensitivity reaction | 0 | 0
  Participants with at least one >= grade 3 rash | 0 | 4

7. Secondary Outcome: Teplizumab Serum Concentrations
Description: PK samples were collected prior to dosing except for Day 9 in Course 1. An additional PK sample was collected 45 minutes after infusion on Day 9 in Course 1. Concentration values below Lower Limit of Quantification (2.50 ng/mL) were set to zero for summary statistics. Course 2 day numbers were set relative to the first day of dosing, regardless of normal or modified dosing schedule.
Time Frame: Pre-dose samples collected on Days 1, 4, 9, 12 and 28 for each of the two treatment courses, and one post-dose sample collected on Day 9 during the first treatment course.
Population: The Pharmacokinetic (PK) population includes all randomized participants who received at least one dose of teplizumab with at least one valid pharmacokinetic sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Teplizumab
Number analyzed (Participants) | 217
ng/mL
  Course 1, Day 1: number analyzed (Participants) | 216
  Course 1, Day 1 | 7.4271 (628.114)
  Course 1, Day 4: number analyzed (Participants) | 210
  Course 1, Day 4 | 70.4769 (50.767)
  Course 1, Day 9: number analyzed (Participants) | 206
  Course 1, Day 9 | 250.3928 (44.677)
  Course 1, Day 9 post-dose: number analyzed (Participants) | 59
  Course 1, Day 9 post-dose | 636.4390 (33.171)
  Course 1, Day 12: number analyzed (Participants) | 208
  Course 1, Day 12 | 305.6569 (47.048)
  Course 1, Day 28: number analyzed (Participants) | 186
  Course 1, Day 28 | 25.0317 (79.953)
  Course 2, Day 1: number analyzed (Participants) | 121
  Course 2, Day 1 | 5.5433 (522.457)
  Course 2, Day 4: number analyzed (Participants) | 123
  Course 2, Day 4 | 82.0166 (50.333)
  Course 2, Day 9: number analyzed (Participants) | 119
  Course 2, Day 9 | 145.9498 (75.737)
  Course 2, Day 12: number analyzed (Participants) | 121
  Course 2, Day 12 | 108.2988 (107.776)
  Course 2, Day 28: number analyzed (Participants) | 118
  Course 2, Day 28 | 13.2159 (181.421)

8. Secondary Outcome: Anti-teplizumab Antibody (ADA) Titers After Treatment Courses
Description: Baseline was defined as the most recent value collected prior to the first dose of study drug. Week 26 Day 187 and Weeks 27 and 34 are planned for subjects under the normal dosing schedule. Week 52 Day 369 and Weeks 53, 56, and 60 are planned for subjects under the modified dosing schedule.
Time Frame: Baseline through 78 Week
Population: The Immunogenicity population includes all randomized participants who received at least one dose of teplizumab with at least one valid serum Anti-teplizumab Antibody (ADA) sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Titer
Arm/Group | Teplizumab
Number analyzed (Participants) | 217
Titer
  Baseline: number analyzed (Participants) | 15
  Baseline | 65.81 (182.3)
  Week 2: number analyzed (Participants) | 176
  Week 2 | 177.22 (278.2)
  Week 4: number analyzed (Participants) | 172
  Week 4 | 817.08 (275.0)
  Week 8: number analyzed (Participants) | 172
  Week 8 | 1040.58 (239.1)
  Week 26 Day 182: number analyzed (Participants) | 134
  Week 26 Day 182 | 834.86 (226.1)
  Week 26 Day 187: number analyzed (Participants) | 124
  Week 26 Day 187 | 807.26 (681.6)
  Week 27: number analyzed (Participants) | 167
  Week 27 | 9257.15 (222.3)
  Week 30: number analyzed (Participants) | 169
  Week 30 | 9985.29 (218.7)
  Week 34: number analyzed (Participants) | 162
  Week 34 | 7326.91 (237.0)
  Week 39: number analyzed (Participants) | 170
  Week 39 | 3701.64 (202.8)
  Week 52 Day 364: number analyzed (Participants) | 153
  Week 52 Day 364 | 1398.22 (240.1)
  Week 52 Day 369: number analyzed (Participants) | 11
  Week 52 Day 369 | 308.80 (207.5)
  Week 53: number analyzed (Participants) | 15
  Week 53 | 8043.22 (165.7)
  Week 56: number analyzed (Participants) | 18
  Week 56 | 14221.44 (241.8)
  Week 60: number analyzed (Participants) | 17
  Week 60 | 9040.49 (299.4)
  Week 65: number analyzed (Participants) | 150
  Week 65 | 996.15 (484.4)
  Week 78: number analyzed (Participants) | 140
  Week 78 | 672.13 (332.4)

9. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA) After Treatment Courses
Description: Baseline is defined as the most recent value collected prior to the first dose of study drug. Week 26 Day 187 and Weeks 27 and 34 are planned for subjects under the normal dosing schedule. Week 52 Day 369 and Weeks 53, 56, and 60 are planned for subjects under the modified dosing schedule.
Time Frame: From baseline through Week 78
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Teplizumab
Number analyzed (Participants) | 217
Participants
  Baseline: number analyzed (Participants) | 215
  Baseline: Positive | 15
  Baseline: Negative | 200
  Week 2: number analyzed (Participants) | 207
  Week 2: Positive | 182
  Week 2: Negative | 25
  Week 4: number analyzed (Participants) | 204
  Week 4: Positive | 178
  Week 4: Negative | 26
  Week 8: number analyzed (Participants) | 206
  Week 8: Positive | 175
  Week 8: Negative | 31
  Week 26 Day 182: number analyzed (Participants) | 192
  Week 26 Day 182: Positive | 139
  Week 26 Day 182: Negative | 53
  Week 26 Day 187: number analyzed (Participants) | 170
  Week 26 Day 187: Positive | 130
  Week 26 Day 187: Negative | 40
  Week 27: number analyzed (Participants) | 175
  Week 27: Positive | 167
  Week 27: Negative | 8
  Week 30: number analyzed (Participants) | 176
  Week 30: Positive | 169
  Week 30: Negative | 7
  Week 34: number analyzed (Participants) | 176
  Week 34: Positive | 163
  Week 34: Negative | 13
  Week 39: number analyzed (Participants) | 192
  Week 39: Positive | 170
  Week 39: Negative | 22
  Week 52 Day 364: number analyzed (Participants) | 192
  Week 52 Day 364: Positive | 155
  Week 52 Day 364: Negative | 37
  Week 52 Day 369: number analyzed (Participants) | 15
  Week 52 Day 369: Positive | 11
  Week 52 Day 369: Negative | 4
  Week 53: number analyzed (Participants) | 16
  Week 53: Positive | 15
  Week 53: Negative | 1
  Week 56: number analyzed (Participants) | 19
  Week 56: Positive | 18
  Week 56: Negative | 1
  Week 60: number analyzed (Participants) | 18
  Week 60: Positive | 17
  Week 60: Negative | 1
  Week 65: number analyzed (Participants) | 191
  Week 65: Positive | 153
  Week 65: Negative | 38
  Week 78: number analyzed (Participants) | 191
  Week 78: Positive | 146
  Week 78: Negative | 45

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events = from the first dose of study drug administration through the end of the study, up to 78 weeks
Groups:
- Placebo; Teplizumab: Safety population
Arm/Group | Placebo | Teplizumab
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/217
Serious Adverse Events (participants affected / at risk) | 6/111 | 12/217
Other Adverse Events (participants affected / at risk) | 88/111 | 212/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=111) | Teplizumab (N=217)
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Palpitation (Cardiac disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Device related bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=111) | Teplizumab (N=217)
Hypotension (Vascular disorders) | 10 | 18
Pyrexia (General disorders) | 11 | 53
Fatigue (General disorders) | 15 | 22
Chills (General disorders) | 0 | 19
Cytokine release syndrome (Immune system disorders) | 1 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 20
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 19
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Lymphocyte count decreased (Investigations) | 5 | 73
White blood cell count decreased (Investigations) | 6 | 53
Neutrophil count decreased (Investigations) | 11 | 33
Alanine aminotransferase increased (Investigations) | 0 | 28
Aspartate Aminotransferase increased (Investigations) | 1 | 20
Tachycardia (Cardiac disorders) | 1 | 12
Headache (Nervous system disorders) | 21 | 94
Dizziness (Nervous system disorders) | 5 | 11
Lymphopenia (Blood and lymphatic system disorders) | 0 | 50
Neutropenia (Blood and lymphatic system disorders) | 1 | 28
Leukopenia (Blood and lymphatic system disorders) | 1 | 26
Anaemia (Blood and lymphatic system disorders) | 5 | 13
Nausea (Gastrointestinal disorders) | 21 | 92
Vomiting (Gastrointestinal disorders) | 15 | 68
Abdominal pain (Gastrointestinal disorders) | 9 | 37
Abdominal pain upper (Gastrointestinal disorders) | 12 | 31
Diarrhoea (Gastrointestinal disorders) | 12 | 31
Rash (Skin and subcutaneous tissue disorders) | 5 | 86
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 29
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 17
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 11
Dermatitis (Skin and subcutaneous tissue disorders) | 6 | 9
Erythema (Skin and subcutaneous tissue disorders) | 6 | 7
Proteinuria (Renal and urinary disorders) | 3 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 15
COVID-19 (Infections and infestations) | 26 | 49
Upper respiratory tract infection (Infections and infestations) | 23 | 44
Nasopharyngitis (Infections and infestations) | 14 | 19
Gastroenteritis (Infections and infestations) | 10 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 81 | 151
Decreased appetite (Metabolism and nutrition disorders) | 3 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 14

LIMITATIONS AND CAVEATS:
Enrollment into the study was temporarily suspended due to COronaVIrus Disease of 2019 (COVID-19) pandemic restrictions. Participants who were unable to receive the second 12-day treatment course at 6 months due to COVID-19 pandemic restrictions were given the second course at approximately 12 months (modified dosing schedule).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has right to publish multi-center study results first, then PI may publish/present study results after Sponsor had at least 60 days and up to 105 days to review/comment/obtain intellectual property protection, PI has deleted all sponsor-requested references to confidential information, and PI has considered the Sponsor's proposed revisions in good faith and meets with the Sponsor to discuss/ resolve any disagreements regarding accuracy, data analyses or confidential information.

DOCUMENTS (2):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT03875729/Prot_002.pdf
  • Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03875729/SAP_003.pdf